CLINICAL TRIAL: NCT02732509
Title: Chronic Inflammation and Exercise Responsiveness
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian R. Lanza, Associate Professor of Medicine, Mayo Clinic
Other Study IDs: 16-000437
Record Dates: First submitted 2016-03-22; First posted 2016-04-08 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Lean: Body mass index less than 25 kg/m2
- Overweight/obese: Body mass index 25-45 kg/m2

SUMMARY:
The purpose of this study is to determine how chronic inflammation influences skeletal muscle protein metabolism and metabolic function in humans. The investigators will evaluate acute responsiveness to a single bout of exercise in men and women who are either lean or overweight/obese. The investigators will explore the relationship between circulating inflammatory markers and anabolic, proteomic, and transcriptional responses to acute exercise. The investigators will measure skeletal muscle protein synthesis in the postabsorptive state and in response to a single bout of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* BMI 19-45 kg/m2

Exclusion Criteria:

* Anemia (female subjects hemoglobin of <11 g/dl and male subjects hemoglobin <12 g/dl)
* Active coronary artery disease or history of unstable macrovascular disease (unstable angina, myocardial infarction, stroke, and revascularization of coronary, peripheral or carotid artery within 3 months of recruitment)
* Renal insufficiency/failure (serum creatinine > 1.5mg/dl)
* Oral warfarin group medications or history of blood clotting disorders.
* Pregnancy or breastfeeding
* Alcohol consumption greater than 2 glasses/day or other substance abuse
* Untreated or uncontrolled thyroid disorders
* Debilitating chronic disease (at the discretion of the investigators)

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women between the ages of 30-55 years will be recruited for this study. Fifteen individuals will be lean, defined as a body mass index (BMI) between 19 and 24 kg/m2. Thirty individuals will be overweight/obese, defined as a BMI between 25 and 45 kg/m2.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption rates in mitochondria isolated from skeletal muscles | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Lanza, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Vanderboom P, Zhang X, Hart CR, Kunz HE, Gries KJ, Heppelmann CJ, Liu Y, Dasari S, Lanza IR. Impact of obesity on the molecular response to a single bout of exercise in a preliminary human cohort. Obesity (Silver Spring). 2022 May;30(5):1091-1104. doi: 10.1002/oby.23419. PMID 35470975
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials